CLINICAL TRIAL: NCT03251482
Title: A Randomized, Double-blind, Double-dummy, Multicenter, Adaptive Design, Dose Escalation (Part 1) and Dose-Response (Part 2) Study to Evaluate the Safety and Efficacy of Intravenous JNJ-64179375 Versus Oral Apixaban in Subjects Undergoing Elective Total Knee Replacement Surgery
Brief Title: A Study to Evaluate the Safety and Efficacy of Intravenous JNJ-64179375 Versus Oral Apixaban in Participants Undergoing Elective Total Knee Replacement Surgery
Acronym: TEXT-TKR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108344; 2016-004550-15 (EudraCT Number); 64179375THR2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: VTE Prophylaxis With Anticoagulation After Total Knee Replacement Surgery
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Double Blinded
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- Part 1: Cohort 1 (0.3 mg/kg JNJ-64179375/Apixaban) (Experimental): Participants will receive JNJ-64179375 0.3 milligram per kilogram (mg/kg) intravenously (IV) or JNJ-64179375 placebo (saline) IV infusion as a single dose on Day 1 and matching apixaban placebo or 2.5 mg apixaban, orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 0.3 mg/kg; Drug: Placebo JNJ-64179375; Drug: Apixaban placebo; Drug: Apixaban 2.5 mg
- Part 1: Cohort 2 (0.6 mg/kg JNJ-64179375/Apixaban) (Experimental): Participants will receive JNJ-64179375 0.6 mg/kg IV or JNJ-64179375 placebo (saline) IV infusion as a single dose on Day 1 and matching apixaban placebo or 2.5 mg apixaban, orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 0.6 mg/kg; Drug: Placebo JNJ-64179375; Drug: Apixaban placebo; Drug: Apixaban 2.5 mg
- Part 1: Cohort 3 (1.2 mg/kg JNJ-64179375/Apixaban) (Experimental): Participants will receive JNJ-64179375 1.2 mg/kg IV or JNJ-64179375 placebo (saline) IV infusion as a single dose on Day 1 and matching apixaban placebo or 2.5 mg apixaban, orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 1.2 mg/kg; Drug: Placebo JNJ-64179375; Drug: Apixaban placebo; Drug: Apixaban 2.5 mg
- Part 1: Optional Cohort 4 (JNJ-64179375/Apixaban) (Experimental): Participants will receive JNJ-64179375 Dose to be determined (TBD) based on preliminary data (dose may range from 0.1 to 1.8 mg/kg or any dose from the preceding cohorts) IV or JNJ-64179375 placebo (saline) IV infusion as a single dose on Day 1 and matching apixaban placebo or 2.5 mg apixaban, orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 (Dose to be Determined); Drug: Placebo JNJ-64179375; Drug: Apixaban placebo; Drug: Apixaban 2.5 mg
- Part 1: Optional Cohort 5 (JNJ-64179375/Apixaban) (Experimental): Participants will receive JNJ-64179375 Dose TBD based on preliminary data (dose may range from 0.1 to 1.8 mg/kg or any dose from the preceding cohorts) IV or JNJ-64179375 placebo (saline) IV infusion as a single dose on Day 1 and matching apixaban placebo or 2.5 mg apixaban, orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 (Dose to be Determined); Drug: Placebo JNJ-64179375; Drug: Apixaban placebo; Drug: Apixaban 2.5 mg
- Part 1: Optional Cohort 6 (JNJ-64179375/Apixaban) (Experimental): Participants will receive JNJ-64179375 Dose TBD based on preliminary data (dose may range from 0.1 to 1.8 mg/kg or any dose from the preceding cohorts) IV or JNJ-64179375 placebo (saline) IV infusion as a single dose on Day 1 and matching apixaban placebo or 2.5 mg apixaban, orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 (Dose to be Determined); Drug: Placebo JNJ-64179375; Drug: Apixaban placebo; Drug: Apixaban 2.5 mg
- Part 2: Group A: JNJ-64179375 A mg/kg and apixaban placebo (Experimental): Participants will receive JNJ-64179375 Dose A mg/kg (TBD based on review of data from Part 1) IV as a single dose on Day 1 and apixaban placebo orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 A mg/kg; Drug: Apixaban placebo
- Part 2: Group B: JNJ-64179375 B mg/kg and apixaban placebo (Experimental): Participants will receive JNJ-64179375 Dose B mg/kg (TBD based on review of data from Part 1) IV as a single dose on Day 1 and apixaban placebo orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 B mg/kg; Drug: Apixaban placebo
- Part 2: Group C: JNJ-64179375 C mg/kg and apixaban placebo (Experimental): Participants will receive JNJ-64179375 Dose C mg/kg (TBD based on review of data from Part 1) IV as a single dose on Day 1 and apixaban placebo orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 C mg/kg; Drug: Apixaban placebo
- Part 2: Group D: JNJ-64179375 D mg/kg and apixaban placebo (Experimental): Participants will receive JNJ-64179375 Dose D mg/kg (TBD based on review of data from Part 1) IV as a single dose on Day 1 and apixaban placebo orally twice a day for 10 to 14 days.
  Interventions: Drug: JNJ-64179375 D mg/kg; Drug: Apixaban placebo
- Part 2: Group E: JNJ-64179375 placebo IV and apixaban 2.5 mg (Experimental): Participants will receive JNJ-64179375 placebo (saline) IV as a single dose on Day 1 and apixaban 2.5 mg orally twice a day for 10 to 14 days.
  Interventions: Drug: Placebo JNJ-64179375; Drug: Apixaban 2.5 mg

INTERVENTIONS:
Drug: JNJ-64179375 0.3 mg/kg — JNJ-64179375 0.3 milligram per kilogram (mg/kg) intravenous (IV) infusion as a single dose on Day 1.
  Arms: Part 1: Cohort 1 (0.3 mg/kg JNJ-64179375/Apixaban)
Drug: JNJ-64179375 0.6 mg/kg — JNJ-64179375 0.6 mg/kg IV infusion as a single dose on Day 1.
  Arms: Part 1: Cohort 2 (0.6 mg/kg JNJ-64179375/Apixaban)
Drug: JNJ-64179375 1.2 mg/kg — JNJ-64179375 1.2 mg/kg IV infusion as a single dose on Day 1.
  Arms: Part 1: Cohort 3 (1.2 mg/kg JNJ-64179375/Apixaban)
Drug: JNJ-64179375 (Dose to be Determined) — JNJ-64179375 IV infusion (Dose to be determined) as a single dose on Day 1.
  Arms: Part 1: Optional Cohort 4 (JNJ-64179375/Apixaban); Part 1: Optional Cohort 5 (JNJ-64179375/Apixaban); Part 1: Optional Cohort 6 (JNJ-64179375/Apixaban)
Drug: JNJ-64179375 A mg/kg — JNJ-64179375 Dose A mg/kg IV as a single dose on Day 1.
  Arms: Part 2: Group A: JNJ-64179375 A mg/kg and apixaban placebo
Drug: JNJ-64179375 B mg/kg — JNJ-64179375 Dose B mg/kg IV as a single dose on Day 1.
  Arms: Part 2: Group B: JNJ-64179375 B mg/kg and apixaban placebo
Drug: JNJ-64179375 C mg/kg — JNJ-64179375 Dose C mg/kg IV as a single dose on Day 1.
  Arms: Part 2: Group C: JNJ-64179375 C mg/kg and apixaban placebo
Drug: JNJ-64179375 D mg/kg — JNJ-64179375 Dose D mg/kg IV as a single dose on Day 1.
  Arms: Part 2: Group D: JNJ-64179375 D mg/kg and apixaban placebo
Drug: Placebo JNJ-64179375 — Matching JNJ-64179375 placebo (normal saline) administered as IV infusion as a single dose on Day 1.
  Arms: Part 1: Cohort 1 (0.3 mg/kg JNJ-64179375/Apixaban); Part 1: Cohort 2 (0.6 mg/kg JNJ-64179375/Apixaban); Part 1: Cohort 3 (1.2 mg/kg JNJ-64179375/Apixaban); Part 1: Optional Cohort 4 (JNJ-64179375/Apixaban); Part 1: Optional Cohort 5 (JNJ-64179375/Apixaban); Part 1: Optional Cohort 6 (JNJ-64179375/Apixaban); Part 2: Group E: JNJ-64179375 placebo IV and apixaban 2.5 mg
Drug: Apixaban placebo — Matching apixaban placebo administered orally twice a day for 10 to 14 days.
  Arms: Part 1: Cohort 1 (0.3 mg/kg JNJ-64179375/Apixaban); Part 1: Cohort 2 (0.6 mg/kg JNJ-64179375/Apixaban); Part 1: Cohort 3 (1.2 mg/kg JNJ-64179375/Apixaban); Part 1: Optional Cohort 4 (JNJ-64179375/Apixaban); Part 1: Optional Cohort 5 (JNJ-64179375/Apixaban); Part 1: Optional Cohort 6 (JNJ-64179375/Apixaban); Part 2: Group A: JNJ-64179375 A mg/kg and apixaban placebo; Part 2: Group B: JNJ-64179375 B mg/kg and apixaban placebo; Part 2: Group C: JNJ-64179375 C mg/kg and apixaban placebo; Part 2: Group D: JNJ-64179375 D mg/kg and apixaban placebo
Drug: Apixaban 2.5 mg — Apixaban 2.5 mg administered orally twice a day for 10 to 14 days.
  Arms: Part 1: Cohort 1 (0.3 mg/kg JNJ-64179375/Apixaban); Part 1: Cohort 2 (0.6 mg/kg JNJ-64179375/Apixaban); Part 1: Cohort 3 (1.2 mg/kg JNJ-64179375/Apixaban); Part 1: Optional Cohort 4 (JNJ-64179375/Apixaban); Part 1: Optional Cohort 5 (JNJ-64179375/Apixaban); Part 1: Optional Cohort 6 (JNJ-64179375/Apixaban); Part 2: Group E: JNJ-64179375 placebo IV and apixaban 2.5 mg

SUMMARY:
The primary purpose of Part 1 in this study is to assess the safety and tolerability of JNJ-64179375 for each dose level for dose escalation and any bleeding events (the composite of major, clinically relevant non-major, and minimal bleeding events) for the selection of doses for Part 2. The primary purpose of Part 2 is to assess the efficacy dose response of JNJ-64179375 for the prevention of total venous thromboembolism (VTE) (proximal and/or distal deep vein thrombosis [DVT] [asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic], nonfatal pulmonary embolism [PE], or any death).

DETAILED DESCRIPTION:
This study has 2 parts, dose escalation and dose-response evaluation, and will be conducted in participants undergoing primary unilateral elective Total Knee Replacement (TKR) surgery. Participants will participate in either Part 1 or Part 2 of study only. The study will be conducted in 3 phases: an up to 30-day screening phase before surgery, a 14-day double-blind dosing phase, and a 16-week follow-up phase. Safety evaluations will include monitoring of all nonserious and serious adverse events, clinical laboratory tests, vital signs measurements, and physical examinations. Pharmacokinetics (dense and sparse), pharmacodynamic (PD), health resource utilization, and immunogenicity samples will also be assessed. The total study duration of participant's participation in Part 1 or part 2 after randomization will be approximately 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than or equal to (>=) 40 kg to less than or equal to (<=) 150 kilogram (kg)
* Medically appropriate for postoperative anticoagulant prophylaxis as determined by the investigator
* Has undergone an elective primary unilateral total knee replacement (TKR)
* Before randomization, a woman must not be of childbearing potential defined as postmenopausal (defined as no menses for 12 months without an alternative medical cause) and/ or permanently sterile (include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy)
* Contraceptive use by men should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies

Exclusion Criteria:

* Any condition for which the use of apixaban is not recommended in the opinion of the investigator
* Bilateral, revision or unicompartmental procedure
* Known or suspected hypersensitivity or intolerance to any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human proteins, monoclonal antibodies or antibody fragments, or any of the excipients of JNJ-64179375
* Unable to undergo venography
* Known previous deep vein thrombosis (DVT) in either lower extremity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (103):
- United States (7):
  - Arizona Research Center, Phoenix, Arizona
  - Harbor-UCLA Medical Center, Torrance, California
  - Denver Metro Orthopedics, PC, Englewood, Colorado
  - Florida Research Associates, LLC, DeLand, Florida
  - Avanza research, Pensacola, Florida
  - University Orthopedic and Joint Replacement Center, Tamarac, Florida
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
- Argentina (7):
  - Hospital Italiano de Buenos Aires, Caba
  - Clínica Adventista Belgrano, CABA
  - Hospital San Roque, Córdoba
  - Clínica Chutro, Córdoba
  - Hospital Italiano La Plata, La Plata
  - Sanatorio Britanico de Rosario, Rosario
  - Sanatorio San Miguel, San Miguel
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt
  - ZNA Jan Palfijn, Merksem
- Brazil (9):
  - Universidade Federal de Minas Gerais (UFMG) - Faculdade de Medicina, Belo Horizonte
  - Hospital Sao Francisco de Assis, Belo Horizonte
  - Unicamp - Hospital de Clinicas, Campinas
  - Uniort.e - Hospital de ortopedia, Londrina
  - Irmandade da Santa Casa de Misericórdia de Marília, Marília
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital e Maternidade Dr Christovão da Gama, Santo André
  - Hospital Estadual Mario covas, Santo André
  - Hospital Das Clinicas Da Faculdade De Medicina Da Universidade De Sao Paulo, São Paulo
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment Russe, Rousse
  - Acibadem City Clinic Tokuda Hospital, Sofa
  - Military Medical Academy, Sofia
- Canada (3):
  - Lakeridge Health Ajax, Ajax, Ontario
  - Source Trial Solutions Inc., Kitchener, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
- Italy (8):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Policlinico San Donato, S. Donato Milanese
  - A.O.U. Città della Salute e della Scienza, Torino
  - Ospedale Mauriziano (Torino), Torino
- Japan (10):
  - Matsudo City General Hospital, Chiba
  - Hakodate Goryokaku Hospital, Hakodate
  - Ritsuzankai Iida Hospital, Iida-shi
  - Itami City Hospital, Itami-shi
  - Yonemori Hospital, Kagoshima
  - Bange Kousei General Hospital, Kawanuma-Gun
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Osaka Rosai Hospital, Osaka
  - Tokushima Municipal Hospital, Tokushima
  - Yuaikai Tomishiro Central Hospital, Tomishiro
- Latvia (4):
  - Regional Hospital of Liepaja, Liepāja
  - Riga 2nd Hospital, Riga
  - Hospital of Traumatology and Orthopedics, Riga
  - Vidzemes Hospital, Valmiera
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital, Klaipėda
- Malaysia (5):
  - University Malaya Medical Center, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Miri, Miri
  - Hospital Sibu, Sibu
  - Hospital Sultan Abdul Halim, Sungai Petani
- Poland (10):
  - Klinika Ortopedii i Traumatologii UMB, Bialystok
  - Oddzial Ortopedii i Traumatologii - Szpital Ogolny im. W.Ginela, Grajewo
  - Klinika Ortopedii Gornoslaskie Centrum Medyczne, Katowice
  - Oddzial Ortopedii i Traumatologii Szpital Specjalistyczny im. L.Rydygiera, Krakow
  - SP ZOZ MSWiA w Krakowie Oddzial Urazowo-Ortopedyczny, Krakow
  - CSK UM Klinika Ortopedii, Lodz
  - Oddzial Urazowo-Ortopedyczny Wojewodzki Szpital Specjalistyczny, Lublin
  - Klinika Ortopedii I Traumatologii,Szpital Kliniczny Ortopedyczno-Rehabilitacyjny UM, Poznan
  - Oddzial Ortopedii Specjalistyczny Szpital im. E.Szczeklika, Tarnów
  - Oddzial Chirurgii Urazowej iOrtopedycznej,Wojewodzki Szpital Brodnowski, SPZOZ, Warsaw
- Russia (8):
  - Barnaul Federal Center of Traumatology, Orthopedics and Endoprothesis replacement, Barnaul
  - Russian Ilizarov Scientific Center For Restorative Traumatology And Ortopaedics, Kurgan
  - Moscow City Clinical Hospital #1 n.a. N.I.Pirogov, Moscow
  - Privolzhsky Research Medical University of Ministry of Health of Russian Federation, Nizhny Novgorod
  - St. Petersburg State Medical Institution City Multifunctional Hospital #2, Saint Petersburg
  - Russian Research Institute of Traumatology and Orthopaedics n.a.R.R.Vreden, Saint Petersburg
  - State Healthcare Institution Samara Regional Clinical Hospital named after V.D.Seredavin, Samara
  - Clinical Emergency Hospital n.a. N.V. Solovyev, Yaroslavl
- Spain (8):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. Fund. Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Univ. I Politecni La Fe, Valencia
- Turkey (Türkiye) (7):
  - Ankara Numune Research and Training Hospital, Ankara
  - Dışkapı Yıldırım Beyazıd Training and Research Hospital, Ankara
  - Yıldırım Beyazıt University Yenimahalle Training and Research Hospital, Ankara
  - Yildirim Beyazit University Medical Faculty Ankara Atatürk Research and Training Hospital, Ankara
  - Bakirkoy Training and Research Hospital, Istanbul
  - Umraniye Training and Research Hospital, Istanbul
  - Izmir Tepecik Training and Research Hospital, Izmir
- Ukraine (8):
  - Municipal Institution Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Institute of Spine and JointPathology named after Prof.Sytenko of NationalAcademy of MedicalSciences, Kharkiv
  - Municipal Institution of Health Care 'Kharkiv Regional Clinical Traumatology Hospital', Kharkiv
  - Kyiv Regional Clinical Hospital, Kyiv
  - Communal Institution of Lviv Regional Council 'Lypa Lviv Regional Hospital', Lviv-Vynnyky
  - Vinnytsya Regional Clinical Hospital named after M.I.Pirogov, Vinnytsia
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 parts: Part 1 (Dose- Escalation) and Part 2 (Dose-Response). After completion of Part 1, the sponsor made the decision to not move forward with Part 2 as there was sufficient data to make a determination of efficacy in Part 1. Part 2 was not conducted, hence endpoints for Part 2 are not reported.
Groups:
- JNJ-64179375 0.3 mg/kg and Apixaban Placebo: Participants received a single intravenous (IV) infusion of JNJ-64179375 0.3 milligrams per kilogram (mg/kg) on Day 1 and matching apixaban placebo tablets orally twice daily (BID) for 10 to 14 days.
- JNJ-64179375 0.6 mg/kg and Apixaban Placebo: Participants received a single IV infusion of JNJ-64179375 0.6 mg/kg on Day 1 and matching apixaban placebo tablets orally BID for 10 to 14 days.
- JNJ-64179375 1.2 mg/kg and Apixaban Placebo: Participants received a single IV infusion of JNJ-64179375 1.2 mg/kg on Day 1 and matching apixaban placebo tablets orally BID for 10 to 14 days.
- JNJ-64179375 1.8 mg/kg and Apixaban Placebo: Participants received a single IV infusion of JNJ-64179375 1.8 mg/kg on Day 1 and matching apixaban placebo tablets orally BID for 10 to 14 days.
- Apixaban 2.5 mg and JNJ-64179375 Placebo IV: Participants received a single IV infusion of matching JNJ-64179375 placebo on Day 1 and apixaban 2.5 mg tablet orally BID for 10 to 14 days.
Period: Overall Study
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Started | 39 | 41 | 43 | 122 | 63
Treated | 38 | 40 | 42 | 122 | 63
Completed | 39 | 40 | 43 | 122 | 63
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose (partial or complete) of active study drug (JNJ-64179375 or apixaban).
Groups:
- Total: Total of all reporting groups
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV | Total
Number analyzed (Participants) | 38 | 40 | 42 | 122 | 63 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.53) | 65.8 (8.14) | 66.9 (6.41) | 67.2 (8.84) | 65.1 (7.01) | 66.4 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 35 | 99 | 42 | 222
  Male | 17 | 15 | 7 | 23 | 21 | 83
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 2 | 9 | 5 | 16
  Black | 1 | 0 | 0 | 1 | 1 | 3
  White | 36 | 39 | 39 | 110 | 54 | 278
  Unspecified | 1 | 1 | 1 | 2 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 2 | 4 | 3 | 8 | 10 | 27
  Belgium | 5 | 3 | 3 | 2 | 3 | 16
  Bulgaria | 0 | 0 | 0 | 2 | 0 | 2
  Canada | 0 | 0 | 0 | 3 | 0 | 3
  Italy | 0 | 1 | 0 | 5 | 2 | 8
  Japan | 0 | 0 | 2 | 5 | 5 | 12
  Latvia | 0 | 0 | 0 | 8 | 4 | 12
  Lithuania | 0 | 0 | 3 | 8 | 1 | 12
  Malaysia | 0 | 0 | 0 | 4 | 0 | 4
  Poland | 17 | 9 | 4 | 18 | 12 | 60
  Russian Federation | 0 | 0 | 2 | 9 | 3 | 14
  Spain | 3 | 3 | 3 | 7 | 2 | 18
  Turkey | 1 | 7 | 5 | 8 | 2 | 23
  Ukraine | 0 | 4 | 7 | 20 | 7 | 38
  United States | 10 | 9 | 10 | 15 | 12 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Bleeding Events (Clinical Events Committee [CEC]- Adjudicated)
Description: Number of participants with treatment-emergent bleeding events (BE) (adjudicated by CEC) were reported. Bleeding event was defined as the composite of major, clinically relevant nonmajor (CRNM), and minimal bleeding events assessed through the Day 10 to 14.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 38 | 40 | 42 | 122 | 63
Participants | 2 | 0 | 5 | 1 | 4

2. Primary Outcome: Number of Participants With Total Venous Thromboembolism (VTE) (CEC-adjudicated)
Description: Number of participants with total VTE were reported. Total VTE was defined as the composite of CEC-adjudicated proximal and/or distal deep vein thrombosis (DVT) (asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic), nonfatal pulmonary embolism (PE), or any death assessed through the Day 10 to 14 visit. 1 participant had an asymptomatic distal clot in the non-operated leg which is not counted in the Total VTE and 2 participants had symptomatic proximal clots at the Day 10 to 14 venography and are counted in both the asymptomatic proximal and symptomatic proximal groups.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: Modified Intent-to-treat (mITT) analysis set included all randomized participants with an evaluable venography assessment or a confirmed symptomatic VTE event, or any death adjudicated by CEC.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 30 | 33 | 30 | 97 | 49
Participants | 10 | 9 | 9 | 31 | 6

3. Secondary Outcome: Number of Participants With Composite of Major and CRNM Bleeding Events (CEC-adjudicated)
Description: Number of participants with composite of major and CRNM bleeding events (adjudicated by CEC) were reported. Major Bleeding: Fatal bleeding; Bleeding that is symptomatic and occurs in critical area/organ and/or; Extrasurgical site bleeding causing fall in Hb level of 20 g/L or more, or leading to transfusion of 2 or more units of whole blood or red cells with temporal association within 24-48 hours to bleeding, and/or; Surgical site bleeding that requires second intervention open, arthroscopic, endovascular, or hemarthrosis resulting in prolonged hospitalization or a deep wound infection and/or; Surgical site bleeding that is unexpected and prolonged and/or sufficiently large to cause hemodynamic instability. CRNM bleeding: acute clinically overt bleeding that does not satisfy additional criteria required for bleeding event to be defined as major BE and meets at least 1 of following criteria: Epistaxis, Gastrointestinal bleed, Hematuria, Bruising/ecchymosis, Hemoptysis, Hematoma.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: Safety analysis set included all randomized participants who received at least 1 dose (partial or complete) of active study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 38 | 40 | 42 | 122 | 63
Participants | 1 | 0 | 2 | 1 | 0

4. Secondary Outcome: Number of Participants With Major Bleeding Event (CEC-adjudicated)
Description: Number of participants with major bleeding events (BE) (adjudicated by CEC) were reported. Major Bleeding: Fatal bleeding; Bleeding that is symptomatic and occurs in critical area/organ and/or; Extrasurgical site bleeding causing fall in hemoglobin (Hb) level of 20 grams per liter (g/L) or more, or leading to transfusion of 2 or more units of whole blood or red cells with temporal association within 24-48 hours to bleeding, and/or; Surgical site bleeding that requires second intervention open, arthroscopic, endovascular, or hemarthrosis resulting in prolonged hospitalization or a deep wound infection and/or; Surgical site bleeding that is unexpected and prolonged and/or sufficiently large to cause hemodynamic instability.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 38 | 40 | 42 | 122 | 63
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Relevant Non-major (CRNM) Bleeding Events (CEC-adjudicated)
Description: Number of participants with CRNM bleeding events (adjudicated by CEC) were reported. CRNM bleeding was defined as acute clinically overt bleeding that does not satisfy additional criteria required for bleeding event to be defined as major bleeding event and meets at least 1 of following criteria: Epistaxis, Gastrointestinal bleed, Hematuria, Bruising/ecchymosis, Hemoptysis, Hematoma.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 38 | 40 | 42 | 122 | 63
Participants | 1 | 0 | 2 | 1 | 0

6. Secondary Outcome: Number of Participants With Major Bleeding or CRNM Bleeding Events (CEC-adjudicated)
Description: Number of participants with major bleeding or CRNM bleeding events (adjudicated by CEC) were reported. Major Bleeding: Fatal bleeding; Bleeding that is symptomatic and occurs in critical area/organ and/or; Extrasurgical site bleeding causing fall in Hb level of 20 g/L or more, or leading to transfusion of 2 or more units of whole blood or red cells with temporal association within 24-48 hours to bleeding, and/or; Surgical site bleeding that requires second intervention open, arthroscopic, endovascular, or hemarthrosis resulting in prolonged hospitalization or a deep wound infection and/or; Surgical site bleeding that is unexpected and prolonged and/or sufficiently large to cause hemodynamic instability. CRNM bleeding: acute clinically overt bleeding that does not satisfy additional criteria required for bleeding event to be defined as major BE and meets at least 1 of following criteria: Epistaxis, Gastrointestinal bleed, Hematuria, Bruising/ecchymosis, Hemoptysis, Hematoma.
Time Frame: Up to Day 10 and 14 (visit observation period)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 38 | 40 | 42 | 122 | 63
Participants | 1 | 0 | 2 | 1 | 0

7. Secondary Outcome: Number of Participants With Minimal Bleeding Events (CEC-adjudicated)
Description: Number of participants with minimal bleeding events (adjudicated by CEC) were reported. Minimal bleeding event was defined as any bleeding event not met major or CRNM criteria.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 38 | 40 | 42 | 122 | 63
Participants | 2 | 0 | 4 | 0 | 4

8. Secondary Outcome: Number of Participants With Major VTE (CEC-adjudicated)
Description: Number of participants with major VTE (adjudicated by CEC) were reported. Major VTE was defined as a composite of proximal DVT (asymptomatic confirmed by venography or objectively confirmed symptomatic), nonfatal PE, or any death. 2 participants had symptomatic proximal clots at the Day 10 to 14 venography and are counted in both the asymptomatic proximal and symptomatic proximal groups.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: mITT analysis set included all randomized participants with an evaluable venography assessment or a confirmed symptomatic VTE event or any death.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 30 | 33 | 30 | 97 | 49
Participants | 2 | 2 | 1 | 7 | 0

9. Secondary Outcome: Number of Participants With Proximal Deep Vein Thrombosis (DVT) (CEC-adjudicated)
Description: Number of participants with proximal DVT (adjudicated by CEC) were reported. DVT asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic. 2 participants had symptomatic proximal clots at the Day 10 to 14 venography and are counted in both the asymptomatic proximal and symptomatic proximal groups.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: mITT analysis set included all randomized participants with an evaluable venography assessment or a confirmed symptomatic VTE event, or any death.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 30 | 33 | 30 | 97 | 49
Participants
  Asymptomatic | 1 | 2 | 0 | 3 | 0
  Symptomatic | 0 | 0 | 0 | 2 | 0

10. Secondary Outcome: Number of Participants With Nonfatal Pulmonary Embolism (PE) (CEC-adjudicated)
Description: Number of participants with nonfatal PE (adjudicated by CEC) were reported.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 30 | 33 | 30 | 97 | 49
Participants | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Death (CEC-adjudicated)
Description: Number of participants with death (adjudicated by CEC) were reported.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 30 | 33 | 30 | 97 | 49
Participants | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Proximal and Distal DVT (CEC-adjudicated)
Description: Number of participants with proximal and distal DVT (adjudicated by CEC) were reported. DVT asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic. 2 participants had symptomatic proximal clots at the Day 10 to 14 venography and are counted in both the asymptomatic proximal and symptomatic proximal groups.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 30 | 33 | 30 | 97 | 49
Participants
  Asymptomatic | 1 | 0 | 1 | 4 | 0
  Symptomatic | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Distal DVT (CEC-adjudicated)
Description: Number of participants with distal DVT (adjudicated by CEC) were reported. DVT asymptomatic confirmed by venography assessment of the operated leg or objectively confirmed symptomatic.
Time Frame: Up to Day 10 to 14 (visit observation period)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
Number analyzed (Participants) | 30 | 33 | 30 | 97 | 49
Participants
  Asymptomatic | 8 | 7 | 8 | 24 | 6
  Symptomatic | 0 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Description: Safety Analysis set included all randomized participants who received at least 1 dose (partial or complete) of active study drug (JNJ-64179375 or apixaban).
Arm/Group | JNJ-64179375 0.3 mg/kg and Apixaban Placebo | JNJ-64179375 0.6 mg/kg and Apixaban Placebo | JNJ-64179375 1.2 mg/kg and Apixaban Placebo | JNJ-64179375 1.8 mg/kg and Apixaban Placebo | Apixaban 2.5 mg and JNJ-64179375 Placebo IV
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40 | 0/42 | 0/122 | 0/63
Serious Adverse Events (participants affected / at risk) | 2/38 | 2/40 | 4/42 | 13/122 | 5/63
Other Adverse Events (participants affected / at risk) | 19/38 | 17/40 | 26/42 | 37/122 | 20/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-64179375 0.3 mg/kg and Apixaban Placebo (N=38) | JNJ-64179375 0.6 mg/kg and Apixaban Placebo (N=40) | JNJ-64179375 1.2 mg/kg and Apixaban Placebo (N=42) | JNJ-64179375 1.8 mg/kg and Apixaban Placebo (N=122) | Apixaban 2.5 mg and JNJ-64179375 Placebo IV (N=63)
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Primary Hyperaldosteronism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Impaired Healing (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Peripheral Swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bladder Cancer Stage 0, with Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bloody Discharge (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 6 | 0
Post Thrombotic Syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-64179375 0.3 mg/kg and Apixaban Placebo (N=38) | JNJ-64179375 0.6 mg/kg and Apixaban Placebo (N=40) | JNJ-64179375 1.2 mg/kg and Apixaban Placebo (N=42) | JNJ-64179375 1.8 mg/kg and Apixaban Placebo (N=122) | Apixaban 2.5 mg and JNJ-64179375 Placebo IV (N=63)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 1
Conjunctival Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 5 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 0
Catheter Site Haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Fat Necrosis (General disorders) | 0 | 1 | 0 | 0 | 0
Feeling Hot (General disorders) | 1 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 2 | 0 | 0
Impaired Healing (General disorders) | 0 | 0 | 1 | 0 | 0
Injection Site Irritation (General disorders) | 1 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 2 | 0
Peripheral Swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 6 | 0 | 0 | 8 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 3 | 1 | 1
Wound Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post Procedural Swelling (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 4 | 2
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Blood Glucose Increased (Investigations) | 1 | 0 | 1 | 1 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Triglycerides Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiovascular Evaluation (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-Glutamyltransferase Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Platelet Count Increased (Investigations) | 0 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1
Dizziness Exertional (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dizziness Postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 3 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Bloody Discharge (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 1 | 0 | 2 | 3
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 4 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Peripheral Venous Disease (Vascular disorders) | 0 | 0 | 0 | 3 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03251482/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT03251482/SAP_001.pdf